CLINICAL TRIAL: NCT03964792
Title: A Phase 1/2 Open Label Study Evaluating the Safety and Efficacy of Gene Therapy of the Sickle Cell Disease by Transplantation of an Autologous CD34+ Enriched Cell Fraction That Contains CD34+ Cells Transduced ex Vivo With the GLOBE1 Lentiviral Vector Expressing the βAS3 Globin Gene (GLOBE1 βAS3 Modified Autologous CD34+ Cells) in Patients With Sickle Cell Disease (SCD)
Brief Title: Safety and Efficacy of Gene Therapy of the Sickle Cell Disease by Transplantation of an Autologous CD34+ Enriched Cell Fraction That Contains CD34+ Cells Transduced ex Vivo With the GLOBE1 Lentiviral Vector Expressing the βAS3 Globin Gene in Patients With Sickle Cell Disease (DREPAGLOBE)
Acronym: DREPAGLOBE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P17006J
Record Dates: First submitted 2019-05-14; First posted 2019-05-28 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DREPAGLOBE drug product (Experimental): The DREPAGLOBE is a genetically modified cell therapy product that consists of autologous human CD34+ hematopoietic stem and progenitor cells (HSPCs) that are enriched in CD34+ cells which have been transduced ex vivo with the lentiviral vector, GLOBE1, expressing an anti-sickling β-globin protein (AS3) containing three amino acid substitutions in the wild-type β-globin gene.
  Interventions: Genetic: DREPAGLOBE drug product

INTERVENTIONS:
Genetic: DREPAGLOBE drug product — Each patient will receive a single IV infusion of DREPAGLOBE drug product

SUMMARY:
The purpose of this study is to evaluate the Safety and Efficacy of Gene Therapy of the Sickle Cell disease by Transplantation of an Autologous CD34+ enriched cell fraction that contains CD34+ cells transduced ex vivo with the GLOBE1 lentiviral vector expressing the βAS3 globin gene (GLOBE1 βAS3 Modified Autologous CD34+ Cells) in Patients with Sickle Cell Disease (SCD)

ELIGIBILITY:
Inclusion Criteria:

* - Age 12-20 years
* Diagnosis of HbSS or S-beta zero thalassemia by Hb electrophoresis or genetic analysis.
* Clinical history or ongoing evidence of severe sickle cell anemia with one OR more of the following clinical complications demonstrating disease severity:

  * At least 3 vaso occlusive crises requiring hospitalization, under hydroxyurea or transfusion, within 2 years prior to enrollment
  * One severe acute chest syndrome (ACS) hospitalized in intensive care unit
  * At least 2 episodes of ACS within the prior 3 years), including one under HU.
  * Acute priapism (at least 2 episodes > 3h in the preceding year or in the year prior to the start of a regular transfusion program), OR stuttering priapism ≥ 1 by week under sickle cell treatment (HU, transfusion or phlebotomy).
  * Cerebral vasculopathy confirmed by MRA (magnetic resonance angiography) without Moya-moya
  * Presence of sickle cell cardiomyopathy documented by Doppler echocardiography (left ventricular ejection fraction (LVEF) <55% AND tricuspid regurgitation velocity >2.5m/s on cardiac echocardiograph),
  * Tricuspid regurgitation velocity >2.8m/s on cardiac echocardiograph without pulmonary hypertension confirmed by right heart catheterization (mPAP<25mmHg)
* Failed hydroxyurea (HU) therapy, were unable to tolerate HU therapy, or, if 18 years of age or older, have actively made the choice to not take the recommended daily HU regimen. Inadequate clinical response to HU, defined as any one of the following outcomes, while on HU for at least 3 months: 2 or more acute sickle pain crises requiring hospitalization, no rise in Hb >1.5 gm/dl from pre-HU baseline or requires transfusion to maintain Hb > 6.0 gm/dL, had an episode of ACS despite adequate supportive care measures.
* Karnovsky/Lansky performance score ≥ 60%
* Sexually active patients must be willing to use an acceptable method of double-barrier contraception for at least 12 months post-infusion (beyond 12 months at the discretion of the investigator)

Exclusion Criteria:

* Chromosomal (karyotyping) or molecular anomalies (detected by NGS) ( ie 7 chromosomal monosomy)
* Existence of a matched sibling donor
* Patients who have started new treatment for SCD within 6months of enrollment
* Hematologic evaluation: Leukopenia (WBC < 3000 µL) ( en cours) or neutropenia (ANC < 1000 µL) or thrombocytopenia (platelet count < 100,000 µL) (not due to an erythropheresis procedure)
* PT/INR or PTT > 1.5 times upper limit of normal (ULN) or clinically significant bleeding disorder
* Evaluations within 6 months prior to screening visit:
* ALT or AST > 3 times ULN
* Liver Cirrhosis suspicion on echography, CT scan or MRI AND confirmed by histology
* Cardiac evaluation: LVEF < 40% by cardiac echocardiogram or by MUGA scan
* Stroke with significant CNS sequelae i.e., Rankin > 2
* Lung interstitial infiltrate AND Forced Vital Capacity less than 70% AND DLCO less than 60% at steady state
* Confirmed pulmonary hypertension defined by a right heart catheterization (PAPm>25mmHg). Right heart catheterization is required if tricuspid regurgitation velocity >2.8m/s on cardiac echocardiograph OR >2.5m/s with an abnormal Brain Natriuretic Peptide dosage or an important decrease in transcutaneous Hb O2 saturation during the 6 minutes walk test.
* Seropositivity for HIV (Human Immunodeficiency Virus), HCV (Hepatitis C Virus), HTLV-1 (Human T-Lymphotropic Virus), or active Hepatitis B Virus, or active infection by CMV or parvovirus B19, based on positive blood PCR.
* Pregnancy or breastfeeding in a postpartum female
* Any current cancer or prior history of a malignant disease, with the exception of curatively treated non-melanoma skin cancer
* Immediate family member with an established or suspected Familial Cancer Syndrome
* Diagnosis of significant psychiatric disorder of the subject that could seriously impeded the ability to participate in the study
* Patients who failed previous HSCT and are severely ill
* Any clinically significant active infection
* Participation in another clinical study with an investigational drug within 30 days of screening
* Any condition, based on perspective of the medical monitor and treating investigator, which may lead to increased safety risk or inability to comply with the protocol

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2019-11-12 (Actual); Primary Completion 2022-07-28 (Actual); Study Completion 2024-01-23 (Actual)

PRIMARY OUTCOMES:
Incidence of transplant related mortality | up to 100 days post treatment
  To evaluate the procedure safety
Incidence of the need for rescue autologous bone marrow transplant | up to 100 days post treatment
  To evaluate the procedure safety
Frequency and severity of AEs post transplant transplant | 6 months post-transplant
  Based on the United States national Cancer Institute Common Terminology Criteria for Adverse Events v4.03 To evaluate the procedure safety
Incidence of vector-derived Replication competent lentivirus (RCL) | 6 months post-transplant
  To evaluate the procedure safety
Incidence of clinically detectable malignancy and/or abnormal clonal dominance assessed as related to study treatment | 6 months post-transplant
  To evaluate the procedure safety.It will be evaluated by vector insertion site analysis (VISA.

SECONDARY OUTCOMES:
Concentration of neutrophil | 6 months post-transplant
  To evaluate the efficacy
Concentration of platelet | 6 months post-transplant
  To evaluate the efficacy. It will be quantified by High performance liquid chromatography
Percentage HbAS3 | 6 months post-transplant
  To evaluate the efficacy. It will be quantified by High performance liquid chromatography It will be quantified by High performance liquid chromatography
Frequency and severity of adverse events | 24 months post-transplant
  based on the United States national Cancer Institute Common Terminology Criteria for Adverse Events v4.03 To evaluate the long -term safety
Absence of RCL (Replication competent lentivirus) | 24 months post-transplant
  To evaluate the long -term safety
Absence of clinically detectable malignancy or abnormal clonal dominance assessed as related to study treatment | 24 months post-transplant
  To evaluate the long -term safety. It will be evaluated by vector insertion site analysis (VISA).
Protein expression through percentage of anti-sickling Hb | 24 months post-transplant
  To evaluate the long -term efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Pablo BARTULOCCI, MD & PhD, Study Director — Department of internal medicine, Henri-Mondor Hospital, Creteil, France.
Locations (1):
- Department of Biotherapy, Necker-Enfants Malades Hospital, Paris, France

REFERENCES:
- [Derived] Sobrino S, Joseph L, Magrin E, Chalumeau A, Hebert N, Corsia A, Denis A, Roudaut C, Aussel C, Leblanc O, Brusson M, Felix T, Diana JS, Petrichenko A, El Etri J, Godard A, Tibi E, Manceau S, Treluyer JM, Mavilio F, Bushman FD, Marcais A, Castelle M, Neven B, Hermine O, Renolleau S, Magnani A, Asnafi V, El Nemer W, Bartolucci P, Six E, Semeraro M, Miccio A, Cavazzana M. Severe inflammation and lineage skewing are associated with poor engraftment of engineered hematopoietic stem cells in patients with sickle cell disease. Nat Commun. 2025 Apr 1;16(1):3137. doi: 10.1038/s41467-025-58321-4. PMID 40169559